CLINICAL TRIAL: NCT03605576
Title: Effect on Symptomatic Release and Sleep Quality of Remote Fu's Subcutaneous Needling on Patients With Chronic Neck Pain
Brief Title: Remote Fu's Subcutaneous Needling for Patients With Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Li-Wei Chou, Minister of Rehabilitation, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH107-REC2-031
Record Dates: First submitted 2018-05-09; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Chronic Neck Pain; Sleep Quality
Keywords: Fu's subcutaneous needle; Transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fu's subcutaneous needling (Experimental): In this arm, the subjects will receive the intervention of FSN on Day1, Day2 and Day4, in total 3 treatments and will be arrange to take efficacy two assessment on Day8 and Day15, separately.
  Interventions: Procedure: Fu's subcutaneous needling
- Transcutaneous electrical nerve stimulation (Active Comparator): In this arm, the subjects will receive the intervention of TENS on Day1, Day2 and Day4, in total 3 treatments and will be arrange to take efficacy two assessment on Day8 and Day15, separately.
  Interventions: Procedure: Transcutaneous electrical nerve stimulation

INTERVENTIONS:
Procedure: Fu's subcutaneous needling — Fu's Subcutaneous Needle (FSN), is an innovation for the treatment of myofascial pain and trigger points. The needle is a non-injection needle, and the fact that both needles are manipulated and act on soft connective tissue.
  FSN abstains from the muscle and deep fascia layers and is confined to only the subcutaneous layer where collagen fibers are most abundant. As the subcutaneous layer is poorly innervated, pain is less than other needling therapies.
  FSN is also currently being used successfully to treat non-musculoskeletal conditions.
  Arms: Fu's subcutaneous needling
Procedure: Transcutaneous electrical nerve stimulation — Transcutaneous electrical nerve stimulation (TENS or TNS) is the use of electric current produced by a device to stimulate the nerves for therapeutic purposes.
  TENS, by definition, covers the complete range of transcutaneously applied currents used for nerve excitation although the term is often used with a more restrictive intent, namely to describe the kind of pulses produced by portable stimulators used to treat pain. The unit is usually connected to the skin using two or more electrodes. A typical batteryoperated TENS unit is able to modulate pulse width, frequency and intensity. Generally TENS is applied at high frequency (>50 Hz) with an intensity below motor contraction (sensory intensity) or low frequency (<10 Hz) with an intensity that produces motor contraction.
  Arms: Transcutaneous electrical nerve stimulation

SUMMARY:
This is a randomized controlled trial to compare the efficacy of Fu's subcutaneous needle (FSN) and Transcutaneous electrical nerve stimulation (TENS) on chronic neck pain by using more objective assessment tools such as Neck Disability Index, Visual Analog Scales, Pressure Pain Threshold and Myotone of MTrPs of Upper Trapezius Muscles, Range of Motion of Stretch of Upper Trapezius Muscle, and Pittsburgh sleep quality index.

DETAILED DESCRIPTION:
Neck pain combining limited range of motion is very common. Lasting for only a few days, it will taper off without any treatment. If the neck pain symptoms persist for more than two months without any improvement, it will be categorized as chronic neck pain causing not only pain but also functional impact, even in daily life, working, and sleep quality.

Fu's subcutaneous needling is utilized in treating disease related with myofascial trigger point, including soft tissue pain, joint pain, even some internal problems. Indeed it reduce pain immediately with no obvious side effects. There were some clinical articles of subjective symptoms description published lacking scientific accessment of efficacy.

Research team leading by Professor Chang-Zern Hong has already prove that excitability can be reduced by distal acupuncture. Needling TE5 and LI11 can reduce pain intensity and average amplitude of MTrPs end plate in upper trapezium m., and increase pain pressure threshold.

Comparing to traditional acupuncture, whether safer and pain-less Fu's subcutaneous needle also has the distal treatment effect or not still needs more scientific experiment to prove. This is a randomized controlled trial to compare the efficacy of Transcutaneous electrical nerve stimulation and Fu's subcutaneous needle on chronic neck pain by using more objective assessment tools such as Neck Disability Index, Visual Analog Scales, Pressure Pain Threshold and Myotone of MTrPs of Upper Trapezius Muscles, Range of Motion of Stretch of Upper Trapezius Muscle, and Pittsburgh sleep quality index.

ELIGIBILITY:
Inclusion Criteria:

* Having chronic neck pain for more than 2 months and subjective subjective pain intensity (VAS) greater than 5 points.
* Patients with myofascial pain diagnosed with unilateral upper trapezius muscle.
* This pain is not effective for previous medication or physical therapy.

Exclusion Criteria:

* Contraindications for general treatment, such as serious medical problems, recent trauma, or pregnancy.
* There has been a history of drug abuse (including excess alcohol) that affects pain assessors.
* Have received neck, upper back, or upper and lower limb surgery.
* People with central or peripheral nerve disease.
* Cognitive dysfunction cannot be matched with the experimenter.
* People with cardiac pacemakers, epilepsy, etc. cannot place electrode patches on the skin.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-04-12 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scales | 1 day
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.

SECONDARY OUTCOMES:
Neck Disability Index | 1 week
  The NDI is a modification of the Oswestry Low Back Pain Disability Index . It is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. The NDI has sufficient support and usefulness to retain its current status as the most commonly used self-report measure for neck pain
Pressure Pain Threshold | 1day
  Pressure pain threshold (PPT) is defined as the minimum force applied which induces pain. This measure has proven to be commonly useful in evaluating tenderness symptom.
Myotone of MTrPs | 1day
  Muscle tone is the muscle's resistance to passive stretch during resting state. Myotone will help the investigators to get muscle parameters such as tone, elasticity and stiffness.
Pittsburgh sleep quality index | 1 week
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete. Developed by researchers at the University of Pittsburgh, the PSQI is intended to be a standardized sleep questionnaire for clinicians and researchers to use with ease and is used for multiple populations. The questionnaire has been used in many settings, including research and clinical activities, and has been used in the diagnosis of sleep disorders. Clinical studies have found the PSQI to be reliable and valid in the assessment of sleep problems to some degree, but more so with self-reported sleep problems and depression-related symptoms than actigraphic measures

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Chou, PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang CH, Tsai LH, Sun MF, Fu Z, Sun J, Chou LW. Rapid Improvement in Neck Disability, Mobility, and Sleep Quality with Chronic Neck Pain Treated by Fu's Subcutaneous Needling: A Randomized Control Study. Pain Res Manag. 2022 Sep 30;2022:7592873. doi: 10.1155/2022/7592873. eCollection 2022. PMID 36247101